CLINICAL TRIAL: NCT00807599
Title: A Phase II Clinical Trial for Untreated Patients With Multiple Myeloma Eligible for Stem Cell Transplant: Lenalidomide (Revlimid®) Plus Low-dose Dexamethasone (Ld x 4 Cycles) Then Stem Cell Collection Followed by Randomization to Continued Ld or Stem Cell Transplantation (SCT) Plus Maintenance L
Brief Title: Lenalidomide (Revlimid®) Plus Low-dose Dexamethasone (Ld x 4 Cycles) Then Stem Cell Collection Followed by Randomization to Continued Ld or Stem Cell Transplantation (SCT) Plus Maintenance L
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Collaborators: Tufts Medical Center (Other); Lahey Clinic (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 08-121
Record Dates: First submitted 2008-12-11; First posted 2008-12-12 (Estimated); Results first posted 2019-03-15 (Actual); Last update posted 2019-03-15 (Actual); Status verified 2018-08

CONDITIONS: Multiple Myeloma
Keywords: CYCLOPHOSPHAMIDE (CYTOXAN); DEXAMETHASONE; G-CSF; Lenalidomide; MELPHALAN; PEG-FILGRASTIM (NEULASTA); 08-121
MeSH Terms: conditions — Multiple Myeloma | interventions — Drug Tapering; Aging; Lenalidomide; Dexamethasone; Drug Tolerance; Therapeutics

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Stem cell transplant x 1 or x 2 (Experimental): All patients on this study start with the same treatment, lenalidomide and dexamethasone by mouth. After patients have received 4 cycles of lenalidomide and dexamethasone and are within 2 weeks of completing stem cell collection, they are randomized (like the toss of a coin) to either :
  * stem cell transplant right after collection
  * continue lenalidomide and dexamethasone, saving stem cell transplant for a later time.
  Interventions: Procedure: Stem cell transplant x 1 or x 2
- Continue lenalidomide and dexamethasone (Experimental): All patients on this study start with the same treatment, lenalidomide and dexamethasone by mouth. After patients have received 4 cycles of lenalidomide and dexamethasone and are within 2 weeks of completing stem cell collection, they are randomized (like the toss of a coin) to either :
  stem cell transplant right after collection
  * continue lenalidomide and dexamethasone
  * saving stem cell transplant for a later time.
  Interventions: Drug: lenalidomide and dexamethasone

INTERVENTIONS:
Procedure: Stem cell transplant x 1 or x 2 — After 4 cycles of Ld, eligible patients will undergo stem cell mobilization and collection with standard-of-care cyclophosphamide and Neupogen (G-CSF) or with plerixafor G-CSF. Mobilization with cyclophosphamide is preferred, but plerixafor is also allowed. Ld will be held for at least 2 weeks prior to stem cell mobilization.
  On the SCT arm, patients not achieving VGPR by 3 months after the 1st SCT will undergo a 2nd SCT. All patients, after one or two SCT, will receive maintenance L.
  Other Names: In the initial 4 cycles of therapy, pts will receive oral lenalidomide at the; starting dose of 25mg on days 1-21 every 28 days (1 cycle) with dose; adjustments for creatinine clearance (CRCL) & dose reductions for toxicity.; Pts will receive low-dose oral dexamethasone at 40mg weekly on days 1, 8, 15 &; 22 of each 28-day cycle with dose reductions as below for toxicity (the weekly; dose could be split over 2 days in the week i.e. 20mg on days 1, 4, 8, 11, 15,; 18, 22, & 25 for better tolerance). For SCT, pts are adm to hosp. High-dose; melphalan is admin in a single dose on day -2 or split dose on days -3 & -2,; through a cvc. Melphalan doseadjustments are made for age & CRCL,. Pts with; CRCL,> 51ml/min receive melphalan at 200mg/m2. Pts with CRCL < 51ml/min; (to be evaluated within 2 weeks of SCT) will receive 140mg/m2. Pts > 70 years; old receive 140mg/m2 also. Each SCT in a tandem SCT is a clinically discrete; event & these rules of dose adjustment apply to each SCT. It is possible,; that pts will get different doses of melphalan in tandem SCT
  Arms: Stem cell transplant x 1 or x 2
Drug: lenalidomide and dexamethasone — Patients will then be randomized to continued Ld or high-dose melphalan with SCT. On the SCT arm patients not achieving VGPR by 3 months after the 1st SCT will undergo a 2nd SCT. All patients after one or two SCT, will receive maintenance L.
  Other Names: In the initial 4 cycles of therapy, pts will receive oral lenalidomide at the; starting dose of 25mg on days 1-21 every 28 days (one cycle) with dose; adjustments for creatinine clearance and dose reductions. Pts will receive; low-dose oral dexamethasone at 40mg weekly on days 1, 8, 15 & 22 of each; 28-day cycle with dose reductions (the weekly dose could be split over 2 days; in the week i.e. 20mg on days 1, 4, 8, 11, 15, 18, 22, & 25 for better; tolerance). For continued Ld, pts will resume Ld at the last dose tolerated; during the initial 4 cycles, with prophylactics & dose reductions as indicated.; Lenalidomide will be continued until progression of disease, if as tolerated.; Low-dose dexamethasone will be continued for 1 year (from the start of initial; treatment), as tolerated. Dose adjustments will follow guidelines. Pts will; be seen every 3 months by their physician & their disease will be reassessed.; Pts will also have a CBC & pregnancy test performed monthly.
  Arms: Continue lenalidomide and dexamethasone

SUMMARY:
The purpose of this study is to compare the effects, good and bad, of two ways to treat patients with standard-risk symptomatic multiple myeloma. Patients with standard-risk myeloma have myeloma with specific features: levels of 2 blood tests have to be in a specific range and there can be no myeloma tumors found outside of the bones or bone marrow, the areas where myeloma is usually discovered. In past clinical studies, patients with standard-risk myeloma have done well with intensive therapy in the form of stem cell transplant. But multiple myeloma is not curable and, although it may respond to standard treatments including stem cell transplant, myeloma always recurs.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 and ≤ 75
* Histologic and serologic findings from MSKCC confirming the diagnosis of multiple myeloma. Standard diagnostic criteria for multiple myeloma will be used, as per the revised International Myeloma Working Group diagnostic criteria.
* Patients must have symptomatic multiple myeloma without advanced organ damage (such as multiple fractures or advanced bone disease causing immobilization, renal failure, spinal cord compression, or organ compromise due to soft tissue plasmacytoma). If immediate therapy with radiation and high-dose steroids (eg, for cord compression) or with bortezomib-based therapy (eg, for renal failure) is required, the patient is not eligible for this trial.
* Patients may have received 1 cycle of prior therapy with dexamethasone for multiple myeloma.
* Adequate organ function is required, defined as follows:
* ANC ≥ 1,500/μl and platelets ≥ 100,000/μl (unless low ANC and platelets are due to multiple myeloma)
* Serum bilirubin ≤ 2.0 mg/dl
* AST, ALT and alkaline phosphatase < 3 times the upper limit of laboratory normal
* Adequate renal function as assessed by calculated creatinine using Cockcroft-Gault estimation of CrCl (see Appendix I): Subjects must have calculated creatinine clearance ≥ 30ml/min by Cockcroft-Gault formula
* Performance status (ECOG) ≤ 2 (Appendix E).
* Eligible for SCT with LVEF ≥ 50% by MUGA or ECHO, and diffusing capacity > 50% predicted by pulmonary function testing
* Ability to understand the investigational nature of this study and to give informed consent
* All study participants must be registered into the mandatory Revlimid REMS® program, and be willing and able to comply with the requirements the of Revlimid REMS® program
* Females of childbearing potential (FCBP)† must have a negative serum or urine pregnancy test with a sensitivity of at least 50 mIU/mL within 10 - 14 days prior to and again within 24 hours prior to prescribing lenalidomide for cycle 1 (prescriptions must be filled within 7 days) and must either commit to continued abstinence from heterosexual intercourse or begin TWO acceptable methods of birth control, one highly effective method and one additional effective method AT THE SAME TIME, at least 28 days before she starts taking lenalidomide. FCBP must also agree to ongoing pregnancy testing. Men must agree not to father a child and agree to use a latex condom during sexual contact with females of child bearing potential even if they have had a successful vasectomy. See Appendix C: Risks of Fetal Exposure, Pregnancy Testing Guidelines and Acceptable Birth Control Methods.
* Able to take aspirin 325mg or 81mg daily as prophylactic anticoagulation (patients intolerant to ASA may use Coumadin or low molecular weight heparin).

Exclusion Criteria:

* Prior treatment for myeloma except for one cycle of dexamethasone
* History of thromboembolic disease within the past 6 months regardless of anticoagulation
* Myocardial infarction within 6 months prior to enrollment, or New York Hospital Association (NYHA) Class III or IV heart failure (see APPENDIX F), uncontrolled angina, severe uncontrolled ventricular arrhythmias, electrocardiographic evidence of acute ischemia or active conduction system abnormalities.
* Pregnant or breast-feeding women are excluded due to the potential teratogenicity of lenalidomide.
* Concurrent active malignancy other than non-melanoma skin cancers or carcinoma-insitu of the cervix, or presence of myelodysplastic or myeloproliferative disease. Patients with prior malignancies with a disease-free interval of ≥ 5 years are eligible.
* Patients who have had prior malignancies within the past 5 years but are considered to be "cured" with a low likelihood of recurrence may be eligible at the discretion of the Principal Investigator.
* Active hepatitis B or C infection
* HIV 1 or 2 positivity
* Any other medical condition or laboratory evaluation that, in the treating physician's or principal investigator's opinion, makes the patient unsuitable to participate in this clinical trial

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 67 (Actual)
Dates: Start 2008-12-10; Primary Completion 2018-07 (Actual); Study Completion 2018-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Hani Hassoun, MD, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (7):
- United States (7):
  - Memoral Sloan Kettering Cancer Center, Basking Ridge, New Jersey
  - Memorial Sloan-Kettering Cancer Center @ Suffolk, Commack, New York
  - Memorial Sloan Kettering West Harrison, Harrison, New York
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - Memorial Sloan Kettering at Mercy Medical Center, Rockville Centre, New York
  - Memoral Sloan Kettering Cancer Center at Phelps, Sleepy Hollow, New York
  - Memorial Sloan Kettering Cancer Center at Phelps Memorial Hospital Center, Sleepy Hollow, New York

REFERENCES:
- See also: Memorial Sloan Kettering Cancer Center — http://www.mskcc.org

RESULTS

PARTICIPANT FLOW:
Groups:
- Continue Lenalidomide and Dexamethasone: All patients on this study start with the same treatment, lenalidomide and dexamethasone by mouth. After patients have received 4 cycles of lenalidomide and dexamethasone and are within 2 weeks of completing stem cell collection, they are randomized (like the toss of a coin) to either :
  stem cell transplant right after collection
  * continue lenalidomide and dexamethasone
  * saving stem cell transplant for a later time.
  lenalidomide and dexamethasone: Patients will then be randomized to continued Ld or high-dose melphalan with SCT. On the SCT arm patients not achieving VGPR by 3 months after the 1st SCT will undergo a 2nd SCT. All patients after one or two SCT, will receive maintenance L.
- Stem Cell Transplant x 1 or x 2: All patients on this study start with the same treatment, lenalidomide and dexamethasone by mouth. After patients have received 4 cycles of lenalidomide and dexamethasone and are within 2 weeks of completing stem cell collection, they are randomized (like the toss of a coin) to either :
  * stem cell transplant right after collection
  * continue lenalidomide and dexamethasone, saving stem cell transplant for a later time.
  Stem cell transplant x 1 or x 2: After 4 cycles of Ld, eligible patients will undergo stem cell mobilization and collection with standard-of-care cyclophosphamide and Neupogen (G-CSF) or with plerixafor G-CSF. Mobilization with cyclophosphamide is preferred, but plerixafor is also allowed. Ld will be held for at least 2 weeks prior to stem cell mobilization.
  On the SCT arm, patients not achieving VGPR by 3 months after the 1st SCT will undergo a 2nd SCT. All patients, after one or two SCT, will receive maintenance L.
- Not Evaluable: Participants were not randomized and are not evaluable
Period: Overall Study
Arm/Group | Continue Lenalidomide and Dexamethasone | Stem Cell Transplant x 1 or x 2 | Not Evaluable
Started | 26 | 24 | 17
Completed | 26 | 24 | 0
Not Completed | 0 | 0 | 17
Not completed — Not treated on protocol study | 0 | 0 | 2
Not completed — Adverse Event | 0 | 0 | 5
Not completed — Inadequate response to induction | 0 | 0 | 9
Not completed — Withdrawal by Subject | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Continue Lenalidomide and Dexamethasone | Stem Cell Transplant x 1 or x 2 | Total
Number analyzed (Participants) | 26 | 24 | 50
Age, Continuous [Mean (Full Range); unit: years] | 61.3 [47 to 71] | 60.5 [50 to 69] | 60.96 [47 to 71]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 13 | 8 | 21
  Male | 13 | 16 | 29
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 1 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 6 | 3 | 9
  White | 19 | 20 | 39
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 1 | 0 | 1
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 26 | 24 | 50

OUTCOME MEASURES:

1. Primary Outcome: Progression Free Survival (PFS) Rate at 2 Years After Enrollment in Untreated Patients With Multiple Myeloma.
Time Frame: 2 years
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Continue Lenalidomide and Dexamethasone | Stem Cell Transplant x 1 or x 2
Number analyzed (Participants) | 26 | 24
percentage of participants | 84.6 [70.7 to 98.5] | 83.3 [68.4 to 98.2]

2. Secondary Outcome: Number of Participants With VGPR + CR Rate
Description: VGPR/Very Good Partial Response + CR/Complete Response (>/= VGPR) for each study arm
  Per Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.0) for target lesions and assessed by MRI: Complete Response (CR), Disappearance of all target lesions; Partial Response (PR), >=30% decrease in the sum of the longest diameter of target lesions; Overall Response (OR) = CR + PR
Time Frame: 2 years
Measure: Count of Participants; unit: Participants
Arm/Group | Continue Lenalidomide and Dexamethasone | Stem Cell Transplant x 1 or x 2
Number analyzed (Participants) | 26 | 24
Participants
  >/= VGPR | 18 | 21
  <VGPR | 8 | 3

3. Secondary Outcome: Overall Response Rates
Description: Per Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.0) for target lesions and assessed by MRI: Complete Response (CR), Disappearance of all target lesions; Partial Response (PR), >=30% decrease in the sum of the longest diameter of target lesions; Overall Response (OR) = CR + PR
Time Frame: 2 years
Measure: Count of Participants; unit: Participants
Arm/Group | Continue Lenalidomide and Dexamethasone | Stem Cell Transplant x 1 or x 2
Number analyzed (Participants) | 26 | 24
Participants
  Stringent Complete Response | 12 | 12
  Very Good Partial Response | 6 | 7
  Partial Response | 8 | 3
  Complete Response | 0 | 2

4. Secondary Outcome: Overall Survival
Time Frame: up to 4 years
Measure: Number (95% Confidence Interval); unit: percentage of participants alive
Arm/Group | Continue Lenalidomide and Dexamethasone | Stem Cell Transplant x 1 or x 2
Number analyzed (Participants) | 26 | 24
percentage of participants alive | 95.7 [87.3 to 99.9] | 90.6 [78.2 to 99.9]

ADVERSE EVENTS:
Time Frame: Up to 4 years
Arm/Group | Continue Lenalidomide and Dexamethasone | Stem Cell Transplant x 1 or x 2
All-Cause Mortality (participants affected / at risk) | 3/26 | 5/24
Serious Adverse Events (participants affected / at risk) | 17/26 | 18/24
Other Adverse Events (participants affected / at risk) | 26/26 | 24/24
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Continue Lenalidomide and Dexamethasone (N=26) | Stem Cell Transplant x 1 or x 2 (N=24)
Arthritis (Musculoskeletal and connective tissue disorders) | 1 | 1
Back Pain (Musculoskeletal and connective tissue disorders) | 2 | 1
Blood Glucose Increase (Metabolism and nutrition disorders) | 1 | 1
Cardiac disorder (Cardiac disorders) | 1 | 0
Cardiac Valve Disease (Cardiac disorders) | 0 | 1
Catheter related infection (Infections and infestations) | 1 | 1
Chest pain (Cardiac disorders) | 1 | 1
Cholecystitis (Hepatobiliary disorders) | 1 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Decubitus ulcer (Skin and subcutaneous tissue disorders) | 1 | 0
Febrile neutropenia (Blood and lymphatic system disorders) | 4 | 4
Hemoglobin decreased (Blood and lymphatic system disorders) | 1 | 2
Infection (Infections and infestations) | 1 | 6
Myelodysplasia (Blood and lymphatic system disorders) | 1 | 0
Myocardial ischemia (Cardiac disorders) | 1 | 1
Neutrophil count decreased (Investigations) | 3 | 1
Osteonecrosis (Musculoskeletal and connective tissue disorders) | 1 | 0
Pain (General disorders) | 1 | 0
Peripheral ischemia (Vascular disorders) | 1 | 0
Pneumonia (Infections and infestations) | 1 | 4
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Rash desquamating (Skin and subcutaneous tissue disorders) | 1 | 0
Respiratory disorder (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Serum sodium decrease (Metabolism and nutrition disorders) | 1 | 0
Soft tissue necrosis lower limb (Musculoskeletal and connective tissue disorders) | 1 | 0
Syncope (Nervous system disorders) | 1 | 1
Thrombosis (Vascular disorders) | 2 | 2
Treatment related secondary malignancy (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 5 | 6
Bronchospasm (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Colitis (Gastrointestinal disorders) | 0 | 1
Confusion (Psychiatric disorders) | 0 | 1
Dehydration (Metabolism and nutrition disorders) | 0 | 1
Diarrhea (Gastrointestinal disorders) | 0 | 1
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Flu-like symptoms (General disorders) | 0 | 1
INR increased (Investigations) | 0 | 1
Joint pain (Musculoskeletal and connective tissue disorders) | 0 | 1
Mental Status (General disorders) | 0 | 1
Muscle weakness (Musculoskeletal and connective tissue disorders) | 0 | 1
Muscle weakness lower limb (Musculoskeletal and connective tissue disorders) | 0 | 1
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 1
Renal failure (Renal and urinary disorders) | 0 | 1
Skin disorder (Skin and subcutaneous tissue disorders) | 0 | 1
Skin infection (Infections and infestations) | 0 | 1
Visceral arterial ischemia (Gastrointestinal disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Continue Lenalidomide and Dexamethasone (N=26) | Stem Cell Transplant x 1 or x 2 (N=24)
ALT (Investigations) | 3 | 9
AST (Investigations) | 3 | 5
Alkaline Phosphatase (Investigations) | 1 | 3
Bilirubin (Investigations) | 3 | 3
CPK (Investigations) | 3 | 1
Constipation (Gastrointestinal disorders) | 3 | 2
Creatinine (Investigations) | 4 | 1
Diarrhea (Gastrointestinal disorders) | 3 | 4
Edema: limb (General disorders) | 2 | 0
Fatigue (General disorders) | 9 | 10
Hyperglycemia (Metabolism and nutrition disorders) | 17 | 13
Hypoglycemia (Metabolism and nutrition disorders) | 2 | 1
Anemia (Blood and lymphatic system disorders) | 20 | 19
INR (Investigations) | 4 | 3
Infection, other (Infections and infestations) | 1 | 5
White Blood Cell (Investigations) | 23 | 22
Lymphopenia (Investigations) | 23 | 22
Magnesium (Metabolism and nutrition disorders) | 3 | 0
Neuropathy: Sensory (Nervous system disorders) | 4 | 4
Neutrophils/Granulocytes (Investigations) | 24 | 21
Headache (Nervous system disorders) | 2 | 0
Pain - Joint (Musculoskeletal and connective tissue disorders) | 3 | 2
Pain, Other (General disorders) | 8 | 6
Hypophosphatemia (Metabolism and nutrition disorders) | 15 | 17
Platelets (Investigations) | 17 | 21
Hyperkalemia (Metabolism and nutrition disorders) | 5 | 2
Hypokalemia (Metabolism and nutrition disorders) | 1 | 7
Rash Desquamation (Skin and subcutaneous tissue disorders) | 2 | 0
Hyponatremia (Metabolism and nutrition disorders) | 4 | 3
Hypoalbuminemia (Metabolism and nutrition disorders) | 0 | 6
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 0 | 3
Febrile Neuropenia (Blood and lymphatic system disorders) | 0 | 2
Fever (General disorders) | 0 | 4
Pain - Pelvis (Reproductive system and breast disorders) | 0 | 2
Pruritus (Skin and subcutaneous tissue disorders) | 0 | 2
Blurred Vision (Eye disorders) | 0 | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-02-13): https://cdn.clinicaltrials.gov/large-docs/99/NCT00807599/Prot_SAP_000.pdf